CLINICAL TRIAL: NCT01883778
Title: Do Providers and Consumers Know the Cost of Common Tests and Procedures Delivered in the Emergency Department?
Brief Title: Evaluating Patient and Physician Cost Knowledge in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Camille Hollifield, PhD, MPH, University of Utah
Other Study IDs: 00057136
Record Dates: First submitted 2013-06-10; First posted 2013-06-21 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Economic Problems
Keywords: Attitudes of health personnel; Attitudes of patients; Medical compliance; Cost awareness; Cost analysis; Patient knowledge; Physician knowledge; Medical economics; Policy; Questionnaires; Health literacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Emergency Department Patients
- Emergency Medicine Physicians

SUMMARY:
The purpose of this study is to identify existing cost knowledge of Emergency Medicine (EM) physicians and patients and investigates its reported impacts on medical compliance. A cross-sectional survey will be administered electronically to Emergency Medicine physicians at the University of Utah Hospital and the Emergency Physician Integrated Care, LLC (EPIC) who staff ten-community hospital Emergency Departments (ED) in order to investigate physician knowledge and attitudes regarding cost and perceived patient compliance. In addition, a cross-sectional survey will be administered to a convenience sample of patients presenting to the University of Utah Emergency Department to obtain information about their cost knowledge and reported compliance. All ED patients will complete a follow-up phone survey to measure compliance with recommendations made during the ED visits. Following administration of the baseline survey physicians will be provided the prices of the test and procedures and will be re-surveyed 30-days later as a post intervention test to measure changes in knowledge and attitudes.

ELIGIBILITY:
Inclusion Criteria Patient Population:

* 18 years old or older
* Deemed psychologically and medically stable by the ED care provide
* Speak English

Exclusion Criteria Patient Population:

* Prisoner
* Brought to Emergency Department by Emergency Medical Service

Inclusion Criteria Physician Population:

* Employed in target medical practices

Exclusion Criteria Physician Population:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be two distinct study populations in this study. The first population will consist of physicians from Emergency Medicine. There are 51 Emergency Medicine physicians at the University of Utah (27 attending, 24 residents); there are 138 board-certified Emergency Medicine physicians in the EPIC group therefore a projected provider cohort of n=90 (about 50% of 189) is anticipated. The only exclusion criterion for physicians is they do not practice in one of the above-mentioned provider groups.
  The second population will consist of patients presenting to the University Utah Emergency Department who are determined by the attending physicians to be mentally and physically competent to complete the questionnaire (n=450). Included in this cohort are all English speaking patients who are eighteen years of age and older, who are deemed psychologically and medically stable by the ED care provider, are not prisoners, and were not brought in by EMS.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of emergency medicine physician with accurate (+/- 25% of actual cost) cost knowledge of common medical services; influence on testing and prescribing patterns. | 1 year
  Measure the extent of formal education regarding cost of medical services that physicians in the survey population have received and how that impacts knowledge and accuracy; perceived impact on medical compliance among patients.

SECONDARY OUTCOMES:
Proportion of emergency department patients with accurate (+/- 25% actual costs) knowledge of medical service cost; correlation between health literacy and cost knowledge accuracy in patients. | 1 year
  Measure patient health literacy using the REALM-SF (AHRQ) and determine any correlation with cost estimation accuracy and reported impact on medical compliance among patients.

OTHER OUTCOMES:
Efficacy of intervention to improving accuracy in cost estimation in emergency physicians. | 1 year
  Changes in self-reported cost knowledge competency and cost estimation accuracy using the intervention comparing the baseline report at time of enrollment to 30 days post intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Broadwater-Hollifield C, Gren LH, Porucznik CA, Youngquist ST, Sundwall DN, Madsen TE. Emergency physician knowledge of reimbursement rates associated with emergency medical care. Am J Emerg Med. 2014 Jun;32(6):498-506. doi: 10.1016/j.ajem.2014.01.044. Epub 2014 Feb 3. PMID 24657227